CLINICAL TRIAL: NCT01185236
Title: A Single Center, Open Label, Randomized Study to Compare the Effect of Vytorin (Simvastatin/Ezetimibe) 10/20mg Versus Atorvastatin 20mg on ApoB/ApoA1 Ratio in Subjects With Diabetes
Brief Title: Study to Compare the Effect of Vytorin (Simvastatin/Ezetimibe) 10/20mg Versus Atorvastatin 20mg on ApoB/ApoA1 Ratio in Subjects With Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Hyun-Jae Kang, Associate professor, Seoul ntional university hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1007-100-324
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes Mellitus Without Insulin Treatment
Keywords: Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Ezetimibe, Simvastatin Drug Combination; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- simvastatin/ezetimibe (vytorin) group (Experimental): vytorin 10/20mg po once daily for 12weeks
  Interventions: Drug: simvastatin/ezetimibe
- atorvastatin group (Active Comparator): atorvastatin 20mg po once daily for 12weeks
  Interventions: Drug: atorvastatin 20mg

INTERVENTIONS:
Drug: simvastatin/ezetimibe — simvastatin/ezetimibe 10/20mg once daily for 12weeks
  Arms: simvastatin/ezetimibe (vytorin) group
Drug: atorvastatin 20mg — atorvastatin 20mg once daily for 12weeks
  Arms: atorvastatin group

SUMMARY:
A single center, open label, randomized, clinical trial comparing ApoB/ApoA ratio of Vytorin 10/20mg vs atorvastatin 20mg treatment.

DM2 patients will be screened for inclusion criteria. Patients (n=66 in each arm) will be randomized to either Ezetimibe/simvastatin 10/20mg or atorvastatin 20mg after 4 week washout or TLC period. Primary and secondary endpoints will be assessed at week 12.

Primary endpoint:

1) change of ApoB/ApoA ratio at week 12.

Secondary endpoint:

1. Change of lipid parameters (TC, LDL-C, HDL-C, TG, apoB 48) at week 12.
2. Change of HbA1C at week 12.
3. Change of HOMA index at week 12

   - HOMA =[Fasting insulin (mIU/L) × Fasting glucose (mmol/L)] / 22.5
4. Change of hsCRP at week 12
5. Safety assessment

Hypotheses:

* Three months treatment of Vytorin 10/20mg will be superior to atorvastatin 20mg in ApoB/ApoA ratio.
* In DM patients, Ezetimibe/Simvastatin Combination will be well-tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 DM
2. Hypercholesterolemia (baseline screening LDL-C > 100 mg/dL)
3. In case of medication, stable doses of oral hypoglycemic agents for at least three months
4. HbA1c <8.5%
5. Age: 20-80

Exclusion Criteria:

1. Chronic renal failure: creatinine > 3.0 mg/dL
2. Serious liver disease (> x3 LFT UNL)
3. Congestive heart failure
4. Stroke or MI/coronary intervention during the preceding 3 months.
5. CK > x 2.5 UNL
6. Unstable hypo/hyperthyroidism
7. Pregnant/lactating woman, or woman intending to become pregnant
8. Subject with any clinically significant condition or situation, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
change of ApoB/ApoA1 | after 12 weeks' treatment
  change of ApoB/ApoA1

SECONDARY OUTCOMES:
change of lipid profile | 12weeks
  change of total cholesterol, LDL-cholesterol, HDL-cholesterol, Triglyceride, and APO B48
change of HbA1c | 12weeks
  change of HbA1c
change of HOMA index | 12weeks
  HOMA =[Fasting insulin (mIU/L) × Fasting glucose (mmol/L)] / 22.5
change of hsCRP | 12weeks
  change of hsCRP
safety | during 12weeks of treatment
  CK elevation, Liver funtion test abnormality, and muscle realted adverse reactions and symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Kang HJ, Kim HS, Sohn DW, Oh BH, Park YB. Effects of ezetimibe/simvastatin 10/20 mg vs. atorvastatin 20 mg on apolipoprotein B/apolipoprotein A1 in Korean patients with type 2 diabetes mellitus: results of a randomized controlled trial. Am J Cardiovasc Drugs. 2013 Oct;13(5):343-51. doi: 10.1007/s40256-013-0031-6. PMID 23728830